CLINICAL TRIAL: NCT05191121
Title: Improving Upper Extremity Function and Trunk Stability After Cervical Spinal Cord Injury (SCI): A Randomized Controlled Trial of Three Interventions
Brief Title: Improving Upper Extremity Function and Trunk Stability After Cervical Spinal Cord Injury (SCI)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Candace Tefertiller, Executive Director Research and Evaluation, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1847023-1
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cervical Spinal Cord Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FTP Alone (Active Comparator): Functional Task Practice Alone - Participants allocated to this group will complete 40 minutes of training focused on improving functional tasks followed by 10 minutes of functional training/carryover in a relevant environment without functional electrical stimulation (FES).
  Interventions: Behavioral: FTP Alone
- FTP+Con-FES (Active Comparator): Functional Task Practice + Conventional Functional Electrical Stimulation - Participants allocated to this group will complete 40 minutes of training focused on improving functional tasks supplemented with conventional parameter (200µs; 40Hz) functional electrical stimulation (FES). followed by 10 minutes of functional training/carryover in a relevant environment.
  Interventions: Behavioral: FTP+Con-FES
- FTP+WPHF-FES (Active Comparator): Functional Task Practice + Wide Pulse, High Frequency Functional Electrical Stimulation - Participants allocated to this group will complete 40 minutes of training focused on improving functional tasks supplemented with wide pulse, high frequency (1000µs; 100 Hz) functional electrical stimulation (FES) followed by 10 minutes of functional training/carryover in a relevant environment.
  Interventions: Behavioral: FTP+WPHF-FES

INTERVENTIONS:
Behavioral: FTP Alone — Participants will be challenged with training speed, weight, limited therapist support, and context variation (e.g., fine motor activities will vary using objects such as cards, dice, coins).
  Arms: FTP Alone
Behavioral: FTP+Con-FES — Participants will be challenged with training speed, weight, limited therapist support, and context variation (e.g., fine motor activities will vary using objects such as cards, dice, coins). Muscle groups will be stimulated at the same time they would be activated naturally in a pre-injury movement pattern utilizing conventional parameter FES.
  Arms: FTP+Con-FES
Behavioral: FTP+WPHF-FES — Participants will be challenged with training speed, weight, limited therapist support, and context variation (e.g., fine motor activities will vary using objects such as cards, dice, coins). Muscle groups will be stimulated at the same time they would be activated naturally in a pre-injury movement pattern utilizing wide pulse, high frequency parameter FES.
  Arms: FTP+WPHF-FES

SUMMARY:
Ninety-nine individuals meeting the study's inclusion/exclusion criteria will be enrolled in this study. The objective of this study is to evaluate three different therapeutic approaches to synergistically retrain functional movement patterns of the upper extremities in combination with trunk stabilization to promote neurologic and functional recovery after SCI. Each subject will complete 40 sessions of intervention. Subjects will also complete a Baseline Evaluation (week 0), Re-Evaluation (week 4), Post Treatment Evaluation (week 8), and a Follow-Up Evaluation (week 12).

ELIGIBILITY:
Inclusion Criteria:

* History of traumatic SCI
* Less than 5months post SCI
* SCI injury level C1-C8
* SCI categorized as AIS B-D
* Currently receiving inpatient rehabilitation at Craig Hospital
* Passive range of motion (ROM) within functional limits at wrists, shoulders, and elbows
* Demonstrate motor response to electrical stimulation in majority of UE muscle groups below level of injury (tested during screening)
* No complicating physical or cognitive conditions (as determined by their physician) that would preclude safe use of electrical stimulation
* Able to complete study as an outpatient if discharged from inpatient rehabilitation before completing 40 sessions of training

Exclusion Criteria:

* Unstable chronic cardiac or respiratory complaints
* Current or history of UE contracture or skin pressure injuries that might interfere with intervention
* Received Botox injections within the last 3 months
* Pregnant
* Implanted devices including: pacemaker, spinal cord stimulator, ventriculoperitoneal shunt, deep brain stimulator, or intra-thecal pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Capabilities of Upper Extremity Test (CUE-T) | Week 0 to Week 12
  32 item test, each item scored on a 0-4 point scale with total scores ranging from 0-128.

SECONDARY OUTCOMES:
Graded Refined Assessment of Strength, Sensibility, and Prehension (GRASSP) | Week 0, Week 8, and Week 12
  This multimodal test measures sensorimotor and prehension function in three domains important in describing arm and hand function
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Sensory Level | Week 0, Week 8, and Week 12
  The ISNCSCI involves a detailed examination to determine the sensory level for the right and left sides. The sensory level is the most caudal, intact dermatome. Scores range from 0-2. The higher the score the more intact the dermatome is.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Motor Level | Week 0, Week 8, and Week 12
  The ISNCSCI involves a detailed examination to determine motor levels for the right and left sides. The motor level is defined as the lowest key muscle function that has a grade of at least a 3, providing key muscle functions represented by segments above that level are judged to be intact. Scores range from 0-5. The higher the score the more intact the muscle is.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Neurological Level of Injury | Week 0, Week 8, and Week 12
  The ISNCSCI involves a detailed examination to determine the neurological level of injury. The neurological level of injury refers to the most caudal segment of the cord with intact sensation and antigravity muscle function strength, provided that there is normal sensory and motor function rostrally respectively. The neurological level of injury is the most cephalad of the sensory and motor levels.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Sacral Sparing | Week 0, Week 8, and Week 12
  The ISNCSCI involves a detailed examination to determine whether a spinal cord injury is complete or incomplete. If an injury is considered complete there is an absence of voluntary anal contraction, absent sensory scores of S4-5, and absence of deep anal pressure.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Impairment Grade | Week 0, Week 8, and Week 12
  The ISNCSCI involves a detailed examination to determine a spinal cord injury's grade according to the American Spinal Injury Association. Score ranges from A-E. ASIA classification A means spinal injury is considered complete with no sensory or motor function preserved in sacral segments. On the opposite end of the scale an ASIA classification E means 'normal'.
Pinch Force | Week 0, Week 8, and Week 12
  Pinch force will be measured by the Commander Echo Console with the JTech Pinch Dynamometer to quantify finger strength.
Grasp Force | Week 0, Week 8, and Week 12
  Grasp force will be measured by the Commander Echo Console with the JTech Hand Dynamometer to quantify grasp strength.
Modified Functional Reach (MFR) | Week 0, Week 8, and Week 12
  The MFR will be used to measure dynamic trunk stability
Global Rating of Change (GRC) | Week 0, Week 8, and Week 12
  The Global Rating of Change scale assesses perceived change from an intervention. 9 point Likert scale. Higher positive score reflects great improvement
NeuroRecovery Scale (NRS) | Week 0 and Week 4
  The full NRS comprises of 16items. For the purpose of this upper extremity interventional study, only six items will be used that represent a variety of functional upper extremity movement patterns required for ADL management. These scores will be used to guide treatment across all 3 groups. Scores range from 1A-4C. Higher scores reflect greater recovery of spinal cord injury.
Demographic Information | Week 0
  Demographic information will include: age, sex, race/ethnic background, pre-injury education, employment status, marital status, and living situation.
Injury Information | Week 0
  Injury information will include: date of injury, cause of injury, baseline AIS classification, and injury level.

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States